CLINICAL TRIAL: NCT01231516
Title: A Randomized, Double-blind Study of the Safety and Efficacy of GSK1349572 50 mg Once Daily Versus Raltegravir 400 mg Twice Daily, Both Administered With an Investigator-selected Background Regimen Over 48 Weeks in HIV-1 Infected, Integrase Inhibitor-Naïve, Antiretroviral-Experienced Adults
Brief Title: A Study of GSK1349572 Versus Raltegravir (RAL) With Investigator Selected Background Regimen in Antiretroviral-Experienced, Integrase Inhibitor-Naive Adults
Acronym: SAILING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111762; 2009-018001-51 (EudraCT Number)
Record Dates: First submitted 2010-10-21; First posted 2010-11-01 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: ART-experienced; Integrase inhibitor; Raltegravir; GSK1349572; Integrase inhibitor naive
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir; Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1349572 + Raltegravir Placebo (Experimental): Subjects will receive GSK1349572 50mg once daily plus raltegravir placebo twice daily.
  Interventions: Drug: GSK1349572; Drug: Raltegravir Placebo
- Raltegravir + GSK1349572 Placebo (Active Comparator): Subjects will receive raltegravir 400mg twice daily plus GSK1349572 placebo once daily.
  Interventions: Drug: Raltegravir; Drug: GSK1349572 Placebo

INTERVENTIONS:
Drug: GSK1349572 — 50mg once daily
  Arms: GSK1349572 + Raltegravir Placebo
Drug: Raltegravir — 400mg twice daily
  Arms: Raltegravir + GSK1349572 Placebo
Drug: GSK1349572 Placebo — Inactive placebo tablet once daily
  Arms: Raltegravir + GSK1349572 Placebo
Drug: Raltegravir Placebo — Inactive placebo tablet twice daily
  Arms: GSK1349572 + Raltegravir Placebo

SUMMARY:
ING111762 is a 48 week, randomized, double-blind, active-controlled, multicenter, parallel group, non-inferiority study. The study will be conducted in at least 688 HIV-1 infected antiretroviral experienced, integrase-naïve subjects. Subjects will be randomized 1:1 to receive GSK1349572 50 mg once daily or raltegravir (RAL) 400 mg twice daily, each added to an investigator selected background regimen consisting of at least one fully active agent plus no more than one second single agent which may or may not be active. Antiviral activity, safety, pharmacokinetics (PK), and development of viral resistance will be evaluated.

DETAILED DESCRIPTION:
ING111762 is a 48 week, randomized, double-blind, active-controlled, multicenter, parallel group, non-inferiority study. The study will be conducted in at least 688 HIV-1 infected antiretroviral experienced, integrase-naïve subjects. Subjects will be randomized 1:1 to receive GSK1349572 50 mg once daily or raltegravir (RAL) 400 mg twice daily, each added to an investigator selected background regimen consisting of at least one fully active agent plus no more than one second single agent which may or may not be active. Antiviral activity, safety, pharmacokinetics (PK), and development of viral resistance will be evaluated.

Subjects must have documented genotypic or phenotypic resistance to at least one member of each of at least two antiretroviral therapy (ART) drug classes [nucleoside/nucleotide reverse transcriptase inhibitor (N[t]RTI), non-nucleoside reverse transcriptase inhibitor (NNRTI), protease inhibitor (PI), fusion inhibitor (T20), or entry inhibitor (chemokine receptor 5 [CCR5] antagonist)].

The primary analysis will take place after the last subject completes 48 weeks on therapy. An additional data cut and analysis will be conducted after the last subject completes 24 weeks on therapy.

Subjects randomized to GSK1349572 who successfully complete Week 48 will continue to received GSK1349572 until either it is locally available, until they no longer derive clinical benefit, until they meet a protocol-defined reason for discontinuation, or until development of the compound is terminated.

ViiV Healthcare is the sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral therapy (ART)-experienced, Human Immunodeficiency Virus (HIV) -1 infected adults at least 18 years of age.
* Women capable of becoming pregnant must use appropriate contraception during the study (as defined by the protocol).
* HIV-1 infection as documented by HIV-1 RNA >400 copies/mL (c/mL) at Screening and with at least one consecutive HIV-1 RNA >400 c/mL within the four months prior to Screening (unless the Screening HIV-1 RNA is > 1000 c/mL where no additional plasma HIV-1 RNA assessment is needed).
* Have documented resistance (via Screening resistance test) to two or more different classes of antiretroviral agents. For subjects off ART for at least one month, if Screening resistance results provide a fully active agent and do not show two class resistance then historical resistance results from the subject's most recent resistance testing may be used, following consultation with the study virologist and /or medical monitor.
* Integrase inhibitor (INI)-naïve, defined as no prior exposure to any INI (e.g. RAL, elvitegravir, or GSK1349572).
* Able to provide written informed consent prior to Screening.
* French subjects: In France, subjects will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Screening resistance test result indicates no fully active antiviral agents are available for design of the background regimen.
* Subject-virus does not yield results using genotype/phenotype/tropism at Screening (assay data is essential for eligibility determination).
* Women who are breastfeeding.
* Any evidence of an active AIDS-defining condition (except cutaneous Kaposi's sarcoma not requiring systemic therapy or CD4+ <200c/mm3).
* Subjects with moderate to severe hepatic impairment as defined by Child-Pugh classification.
* Recent history (less than or equal to 3 months) of upper or lower gastrointestinal bleed, with the exception of anal or rectal bleeding.
* Anticipated need for hepatitis C therapy during the study.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class.
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma; other localized malignancies require agreement between the investigator and study medical monitor for inclusion of the subject.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days prior to Screening.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, any immunomodulator.
* Treatment with any agent, other than licensed ART, which has documented activity against HIV-1 in vitro within 28 days of first dose of investigational product.
* Exposure to an experimental drug and/or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the experimental test agent - whichever is longer, prior to the first dose of IP.
* French subjects recruited at sites in France will be excluded if the subject has participated in any study using an investigational drug and/or vaccine within 60 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine - whichever is longer - prior to screening for the study or the subject plans to participate simultaneously in another clinical study.
* Any acute or verified Grade 4 laboratory abnormality.
* Alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN).
* ALT greater than or equal to 3xULN and bilirubin greater than or equal to 1.5xULN (with >35% direct bilirubin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2010-10-26 (Actual); Primary Completion 2013-02-04 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (145):
- United States (55):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Wilton Manors, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
- Argentina (5):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Australia (2):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Melbourne, Victoria
- Belgium (4):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Liège
- Brazil (8):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, Santos
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Chile (3):
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- France (8):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Garches
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Tourcoing
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Piraeus
  - GSK Investigational Site, Rio, Patras
- GSK Investigational Site, Budapest, Hungary
- Italy (6):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Busto Arsizio (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
- Mexico (4):
  - GSK Investigational Site, León, Guanajuato, Guanajuato
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuautitlán, Estado de México, State of Mexico
  - GSK Investigational Site, Mexico City
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, Chorzów, Poland
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
- Russia (11):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, N.Novgorod
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Toliyatti
  - GSK Investigational Site, Volgograd
  - GSK Investigational Site, Yekaterinburg
- South Africa (3):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Durban
- Spain (16):
  - GSK Investigational Site, (Móstoles) Madrid
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Granollers (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- United Kingdom (4):
  - GSK Investigational Site, Woolwich, London, London
  - GSK Investigational Site, Crumpsall, Manchester
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Tooting, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Cahn P, Pozniak AL, Mingrone H, Shuldyakov A, Brites C, Andrade-Villanueva JF, Richmond G, Buendia CB, Fourie J, Ramgopal M, Hagins D, Felizarta F, Madruga J, Reuter T, Newman T, Small CB, Lombaard J, Grinsztejn B, Dorey D, Underwood M, Griffith S, Min S; extended SAILING Study Team. Dolutegravir versus raltegravir in antiretroviral-experienced, integrase-inhibitor-naive adults with HIV: week 48 results from the randomised, double-blind, non-inferiority SAILING study. Lancet. 2013 Aug 24;382(9893):700-8. doi: 10.1016/S0140-6736(13)61221-0. Epub 2013 Jul 3. PMID 23830355
- [Derived] Benlarbi M, Richard J, Clemente T, Bourassa C, Tolbert WD, Prakash M, Chandravanshi M, Clark A, Pazgier M, Durand M, Castagna A, Finzi A. Fostemsavir Decreases the Levels of Anti-gp120 CD4-Induced Antibodies in Heavily Treatment-Experienced People With HIV. J Infect Dis. 2025 Sep 24:jiaf461. doi: 10.1093/infdis/jiaf461. Online ahead of print. PMID 40990223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted to demonstrate non-inferior antiviral activity of dolutegravir (DTG) 50 milligram (mg) once daily versus raltegravir (RAL) 400 mg twice daily in participants with human immunodeficiency viruses (HIV)-1. Long-term antiviral activity, tolerability & safety were also evaluated
Pre-assignment Details: 1441 participants screened; 724 participants randomized, of which 5 participants did not receive study treatment. 719 participants received at least 1 dose of study medication creating the intent to treat exposed (ITT-E) Population.
Groups:
- DTG 50 mg OD: Participants received dolutegravir (DTG) 50 milligrams (mg) once daily (OD) + matching Raltegravir (RAL) placebo twice daily (BID), one in the morning (AM dose) and one in the evening (PM dose) + investigator selected background antiretroviral (ART) therapy for 48 weeks. Participants who successfully completed 48 weeks of treatment continued to have access to DTG in the Open-Label phase of the study.
- RAL 400 mg BID: Participants received matching DTG placebo OD + RAL 400 mg BID as AM and PM doses + investigator selected background ART therapy for 48 weeks. Participants were discontinued from the study after completion of the Week 48 visit unless a participant successfully completed Week 48 and RAL was not approved and commercially available within the country, GlaxoSmithKline (GSK) continued to supply RAL in the Open-Label Phase until commercially available.
Period: Double-blind Phase (Up to Week [Wk] 48)
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Started (Randomized) | 360 | 364
ITT-E Population | 357 | 362
Modified (m)ITT-E Population | 354 | 361
Completed | 299 | 283
Not Completed | 61 | 81
Not completed — Adverse Event | 4 | 11
Not completed — Lack of Efficacy | 20 | 42
Not completed — Protocol Violation | 9 | 6
Not completed — Met Protocol-Defined Stopping Criteria | 5 | 3
Not completed — Lost to Follow-up | 5 | 10
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Site Closed | 3 | 1
Not completed — Randomized, but did not receive treatment | 3 | 2
Period: Open-label Phase:From Wk 48 up to Wk 480
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Started | 295 (4 participants completed the Double-blind Phase but did not enter the Open-label Phase.) | 126 (157 participants completed the Double-blind Phase but did not enter the Open-label Phase.)
Completed | 227 | 109
Not Completed | 68 | 17
Not completed — Physician Decision | 5 | 0
Not completed — Lack of Efficacy | 27 | 11
Not completed — Protocol Violation | 10 | 0
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Met protocol-defined stopping criteria | 2 | 0
Not completed — Adverse Event | 6 | 1
Not completed — Lost to Follow-up | 12 | 2

BASELINE CHARACTERISTICS:
Population: Four participants from one closed site were removed from the ITT-E Population creating the modified ITT-E Population with 715 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG 50 mg OD | RAL 400 mg BID | Total
Number analyzed (Participants) | 354 | 361 | 715
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristic data are reported for members of the modified Intent-To-Treat Exposed Population, all randomized participants who received at least one dose of IP excluding four participants at one site, which was closed due to Good Clinical Practice (GCP) non-compliance issues in another ViiV sponsored trial.
  Years | 42.6 (10.45) | 42.5 (9.81) | 42.5 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristic data are reported for members of the modified Intent-To-Treat Exposed Population, all randomized participants who received at least one dose of IP excluding four participants at one site, which was closed due to Good Clinical Practice (GCP) non-compliance issues in another ViiV sponsored trial.
  Participants
    Female | 107 | 123 | 230
    Male | 247 | 238 | 485
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Baseline Characteristic data are reported for members of the modified Intent-To-Treat Exposed Population, all randomized participants who received at least one dose of IP excluding four participants at one site, which was closed due to Good Clinical Practice (GCP) non-compliance issues in another ViiV sponsored trial.
  Participants
    African American/African Heritage | 143 | 160 | 303
    American Indian or Alaska Native | 10 | 17 | 27
    Asian-Central/South Asian Heritage | 2 | 2 | 4
    Asian-East Asian Heritage | 6 | 4 | 10
    Asian-South East Asian Heritage | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    White-Arabic/North African Heritage | 3 | 3 | 6
    White-White/Caucasian/European Heritage | 175 | 172 | 347
    Mixed Race | 12 | 2 | 14
    Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) <50 Copies/Milliliter (c/mL) at Week 48
Description: The percentage of participants with Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) <50 c/mL at Week 48 was assessed using the Missing, Switch or Discontinuation = Failure (MSDF), as codified by the Food and Drug Administration (FDA) "snapshot" algorithm. This algorithm treated all participants without HIV-1 RNA at Week 48 as nonresponders, as well as participants who switched their concomitant ART prior to Week 48 as follows: background ART substitutions non-permitted per protocol (one background ART substitution was permitted for safety or tolerability); background ART substitutions permitted per protocol unless the decision to switch was documented as being before or at the first on-treatment visit where HIV-1 RNA was assessed. Otherwise, virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment in the randomized phase of the study.
Time Frame: At Week 48
Population: Modified Intent-To-Treat Exposed (mITT-E) Population: All randomized participants who received at least one dose of investigational product (IP) excluding four participants at one site, which was closed due to Good Clinical Practice (GCP) non-compliance issues in another ViiV sponsored trial.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Percentage of participants | 71 | 64
Statistical Analysis 1: Comparison: DTG 50 mg OD vs RAL 400 mg BID; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTG 50 mg and RAL at Week 48 can be concluded if the lower bound of a two-sided 95% confidence interval (CI) for the difference in percentages (DTG - RAL) is greater than -12%. If non-inferiority were established, superiority would be tested at the nominal 5% level based on a pre-specified testing procedure; p = 0.030, Cochran-Mantel-Haenszel — P-value is for test of superiority; Adjusted difference in proportion which is based on the difference in percentage, adjusted for Baseline (BL) stratification factors; Difference in percentage = 7.4, 95% CI 2-sided [0.7 to 14.2] — Analysis was adjusted for BL stratification factors: HIV-1 RNA (<=50000 versus [vs]>50000 c/mL), darunavir-ritonavir use without primary protease inhibitor mutations (yes vs no), and phenotypic susceptibility score (2 vs <2) to background regimen

2. Secondary Outcome: Number of Participants (Par.) With Detectable Virus That Has Genotypic or Phenotypic Evidence of Treatment-emergent Integrase Inhibitor (INI) Resistance at Time of Protocol Defined Virology Failure (PDVF)
Description: For par. meeting one of the criteria for PDVF, plasma samples collected at the time point of virologic failure and Baseline were tested to evaluate any potential genotypic and/or phenotypic evolution of resistance. PDVF was defined as (A) virologic non-response: a decrease in plasma HIV-1 RNA of <1 logarithm to base 10 (log10) copies/mL by Week 16, with subsequent confirmation, unless plasma HIV-1 RNA is <400 copies/ mL; confirmed plasma HIV-1 RNA levels >=400 copies/mL on or after Week 24 or (B) virologic rebound: confirmed rebound in plasma HIV-1 RNA levels to >=400 copies/mL after prior confirmed suppression to <400 copies/mL; confirmed plasma HIV-1 RNA levels >1 log10 copies/mL above the nadir value, where nadir is >=400 copies/mL.Treatment-emergent IN mutations are those detected at the time of PDVF but not at Baseline.
Time Frame: Baseline (Day 1) until PDVF (Up to Week 48)
Population: mITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Participants | 4 | 17

3. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 c/mL at Week 24
Description: The number of participants with Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) <50 c/mL at Week 24 was assessed using the Missing, Switch or Discontinuation = Failure (MSDF), as codified by the Food and Drug Administration (FDA) "snapshot" algorithm. This algorithm treated all participants without HIV-1 RNA at Week 24 as nonresponders, as well as participants who switched their concomitant ART prior to Week 24 as follows: background ART substitutions non-permitted per protocol (one background ART substitution was permitted for safety or tolerability); background ART substitutions permitted per protocol unless the decision to switch was documented as being before or at the first on-treatment visit where HIV-1 RNA was assessed. Otherwise, virologic success or failure was determined by the last available HIV-1 RNA measurement through Week 24 (within window) while the participant was on-treatment. The result below corresponds to the Week 24 interim analysis.
Time Frame: At Week 24
Population: mITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Participants | 281 | 252

4. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <400 c/mL at Week 24 and Week 48
Description: The number of participants with Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) <400 c/mL at the visit of interest was assessed using the Missing, Switch or Discontinuation = Failure (MSDF), as codified by the Food and Drug Administration (FDA) "snapshot" algorithm. This algorithm treated all participants without HIV-1 RNA at the visit of interest as nonresponders, as well as participants who switched their concomitant ART prior to the visit of interest as follows: background ART substitutions non-permitted per protocol (one background ART substitution was permitted for safety or tolerability); background ART substitutions permitted per protocol unless the decision to switch was documented as being before or at the first on-treatment visit where HIV-1 RNA was assessed. Otherwise, virologic success or failure was determined by the last available HIV-1 RNA measurment (within window) for the timepoint of interest while the participant was on-treatment.
Time Frame: At Week 24 and Week 48
Population: mITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Participants
  Week 24 | 307 | 287
  Week 48 | 278 | 257

5. Secondary Outcome: Absolute Values of Cluster of Differentiation 4+ (CD4+) Cell Counts at Baseline (Day 1) and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 96 and 144
Description: Blood samples were collected at specified time points to assess CD4+ using flow cytometry. Median and interquartile range are presented. Baseline was the latest pre-dose assessment value (Day 1).
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 96 and 144
Population: mITT-E Population. Only those participants with data available at the specified time points were analyzed (represented by "n=X" in the category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Cells per cubic millimeter
  Baseline (Day 1), n=354, 361 | 204.5 [88 to 368] | 193.0 [96 to 365]
  Week 4, n=341, 351: number analyzed (Participants) | 341 | 351
  Week 4, n=341, 351 | 266.0 [164 to 416] | 253.0 [153 to 425]
  Week 8, n=338, 346: number analyzed (Participants) | 338 | 346
  Week 8, n=338, 346 | 280.0 [179 to 423] | 268.0 [163 to 445]
  Week 12, n=335, 345: number analyzed (Participants) | 335 | 345
  Week 12, n=335, 345 | 296.0 [188 to 451] | 289.0 [174 to 443]
  Week 16, n=327, 338: number analyzed (Participants) | 327 | 338
  Week 16, n=327, 338 | 299.0 [179 to 462] | 293.0 [186 to 460]
  Week 24, n=326, 326: number analyzed (Participants) | 326 | 326
  Week 24, n=326, 326 | 334.5 [201 to 488] | 326.5 [198 to 473]
  Week 32, n=309, 309: number analyzed (Participants) | 309 | 309
  Week 32, n=309, 309 | 332.0 [229 to 482] | 338.0 [215 to 484]
  Week 40, n=299, 292: number analyzed (Participants) | 299 | 292
  Week 40, n=299, 292 | 376.0 [239 to 523] | 349.0 [227 to 500]
  Week 48, n=298, 286: number analyzed (Participants) | 298 | 286
  Week 48, n=298, 286 | 387.0 [247 to 565] | 378.5 [247 to 521]
  Week 96, n=260, 22: number analyzed (Participants) | 260 | 22
  Week 96, n=260, 22 | 436.5 [300 to 616] | 484.5 [393 to 573]
  Week 144, n=192, 18: number analyzed (Participants) | 192 | 18
  Week 144, n=192, 18 | 500.0 [346 to 657] | 535.0 [371 to 579]

6. Secondary Outcome: Change From Baseline in CD4+ Cell Counts at Weeks 4, 8, 12,16, 24, 32, 40, 48, 96 and 144
Description: Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline was the latest pre-dose assessment value (Day 1). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Median and interquartile range is presented.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 24, 32, 40, 48, 96 and 144
Population: mITT-E Population Only those participants with data available at the specified data points were assessed (represented by "n=X" in the category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Cells per cubic millimeter
  Week 4, n=341, 351: number analyzed (Participants) | 341 | 351
  Week 4, n=341, 351 | 53.0 [0 to 109] | 45.0 [5 to 99]
  Week 8, n=338, 346: number analyzed (Participants) | 338 | 346
  Week 8, n=338, 346 | 60.5 [15 to 117] | 59.0 [12 to 124]
  Week 12, n=335, 345: number analyzed (Participants) | 335 | 345
  Week 12, n=335, 345 | 74.0 [25 to 135] | 75.0 [22 to 141]
  Week 16, n=327, 338: number analyzed (Participants) | 327 | 338
  Week 16, n=327, 338 | 76.0 [20 to 156] | 79.5 [28 to 158]
  Week 24, n=326, 326: number analyzed (Participants) | 326 | 326
  Week 24, n=326, 326 | 99.0 [34 to 184] | 93.0 [46 to 166]
  Week 32, n=309, 309: number analyzed (Participants) | 309 | 309
  Week 32, n=309, 309 | 107.0 [49 to 188] | 116.0 [52 to 173]
  Week 40, n=299, 292: number analyzed (Participants) | 299 | 292
  Week 40, n=299, 292 | 125.0 [57 to 212] | 117.5 [51.5 to 192]
  Week 48, n=298, 286: number analyzed (Participants) | 298 | 286
  Week 48, n=298, 286 | 144.0 [73 to 239] | 137.0 [65 to 222]
  Week 96, n=260, 22: number analyzed (Participants) | 260 | 22
  Week 96, n=260, 22 | 198.5 [92.5 to 299.5] | 270 [209 to 348]
  Week 144, n= 192, 18: number analyzed (Participants) | 192 | 18
  Week 144, n= 192, 18 | 243.0 [138 to 357] | 302.5 [154 to 390]

7. Secondary Outcome: Number of Participants With Post-Baseline HIV-associated Conditions, Excluding Recurrences, and Disease Progressions
Description: Clinical disease progression (CDP) was assessed according to the Centers for Disease Control and Prevention (CDC) HIV-1 classification system. Category (CAT) A: one or more of following conditions (CON), without any CON listed in Categories B and C: Asymptomatic HIV infection, persistent generalized lymphadenopathy, acute (primary) HIV infection with accompanying illness or history of acute HIV infection. CAT B: Symptomatic CON that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or that are considered by physicians to have clinical course or to require management that is complicated by HIV infection; and not included among CON listed in clinical CAT C. CAT C:Clinical CON listed in acquired immunodeficiency syndrome (AIDS) surveillance case definition. Indicators of CDP defined as:CDC CAT A at Baseline (BS) to CDC CAT C event (EV); CDC CAT B at BS to CDC CAT C EV; CDC CAT C at BS to new CDC CAT C EV; or CDC CAT A, B, or C at BS to death.
Time Frame: Up to Week 480
Population: mITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Participants
  Any CAT | 32 | 25
  CAT B | 16 | 14
  CAT C | 12 | 8
  Death | 6 | 4
  Progression from CAT A to CAT C | 2 | 1
  Progression from CAT B to CAT C | 0 | 1
  Progression from CAT C to New CAT C | 9 | 5
  Progression from CAT A, B, or C to Death | 6 | 4

8. Secondary Outcome: Number of Participants With Post-Baseline Emergent Grade 1 to 4 Clinical Chemistry and Hematology Toxicities
Description: All Grade 1 to 4 post-Baseline-emergent chemistry toxicities included alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), asparate aminotransferase (AST), carbon dioxide (CO2) content/bicarbonate, cholesterol, creatine kinase (CK), creatinine, hyperglycemia, hyperkalemia, hypernatremia, hypoglycemia, hypokalemia, hyponatremia, low density lipoprotein (LDL) cholesterol calculation, lipase, total bilirubin, and triglycerides. All Grade 1 to 4 post-Baseline-emergent hematology toxities included hemoglobin, platelet count, total neutrophils, and white blood cell count. The Division of AIDS (DAIDS) defined toxicity grades as follows: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening; Grade 5, death. Higher the grade, more severe the symptoms.
Time Frame: From Baseline (Day 1) until Week 48, including participants with post-treatment events occurring after Week 48 for participants not entering the post-Week 48 Open-Label phase of the study
Population: Safety Population comprised of all participants who received at least one dose of IP (i.e., DTG or RAL)
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 357 | 362
Participants
  ALT | 47 | 46
  Albumin | 4 | 3
  ALP | 27 | 42
  AST | 49 | 52
  CO2 content/bicarbonate | 97 | 109
  Cholesterol | 99 | 103
  CK | 28 | 29
  Creatinine | 18 | 13
  Hyperglycaemia | 71 | 80
  Hyperkalemia | 7 | 6
  Hypernatremia | 5 | 7
  Hypoglycaemia | 21 | 14
  Hypokalemia | 37 | 41
  Hyponatremia | 76 | 79
  LDL cholesterol calculation | 68 | 82
  Lipase | 63 | 68
  Total bilirubin | 56 | 53
  Triglycerides | 14 | 24
  Hemoglobin | 19 | 27
  Platelet count | 36 | 32
  Total neutrophils | 49 | 49
  White Blood Cell count | 19 | 29

9. Secondary Outcome: Number of Participants With Post-Baseline Emergent Grade 1 to 4 Clinical Chemistry and Hematology Toxicities
Description: Blood samples were collected for the analysis of clinical chemistry and hematology parameters: Alanine aminotransferase (ALT), albumin, alkaline phosphate (ALP), aspartate aminotransferase (AST), carbon dioxide (CO2) content/bicarbonate, cholesterol, creatine kinase (CK), creatinine, hyperglycemia, hyperkalemia, hypernatremia, hypoglycemia, hypokalemia, hypoonatremia, LDL cholesterol, lipase, total bilirubin, triglycerides, hemoglibin, neutrophils, platelets, white blood cells. Any abnormality in clinical chemistry and hematology parameters were evaluated according to the DAIDS toxicity scale From Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening).Higher the grade, more severe the symptoms.
Time Frame: From Week 48 to Week 480
Population: Safety Population. Only those participants who completed Week 48 and continued into open-label phase were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 295 | 126
Participants
  ALT, Grades 1 to 4 | 36 | 9
  ALT, Grades 2 to 4 | 11 | 3
  ALT, Grades 3 to 4 | 4 | 0
  Albumin, Grades 1 to 4 | 3 | 0
  Albumin, Grades 2 to 4 | 3 | 0
  Albumin, Grades 3 to 4 | 0 | 0
  ALP, Grades 1 to 4 | 20 | 1
  ALP, Grades 2 to 4 | 4 | 1
  ALP, Grades 3 to 4 | 1 | 1
  AST, Grades 1 to 4 | 36 | 8
  AST, Grades 2 to 4 | 14 | 0
  AST, Grades 3 to 4 | 1 | 0
  CO2 content/bicarbonate, Grades 1 to 4 | 100 | 21
  CO2 content/bicarbonate, Grades 2 to 4 | 12 | 3
  CO2 content/bicarbonate, Grades 3 to 4 | 0 | 0
  Cholesterol, Grades 1 to 4 | 138 | 26
  Cholesterol, Grades 2 to 4 | 66 | 16
  Cholesterol, Grades 3 to 4 | 11 | 3
  CK, Grades 1 to 4 | 35 | 4
  CK, Grades 2 to 4 | 11 | 1
  CK, Grades 3 to 4 | 2 | 1
  Creatinine, Grades 1 to 4 | 20 | 2
  Creatinine, Grades 2 to 4 | 8 | 2
  Creatinine, Grades 3 to 4 | 2 | 1
  Hyperglycemia, Grades 1 to 4 | 94 | 10
  Hyperglycemia, Grades 2 to 4 | 40 | 6
  Hyperglycemia, Grades 3 to 4 | 7 | 1
  Hyperkalemia, Grades 1 to 4 | 9 | 1
  Hyperkalemia, Grades 2 to 4 | 4 | 1
  Hyperkalemia, Grades 3 to 4 | 2 | 0
  Hypernatremia, Grades 1 to 4 | 7 | 1
  Hypernatremia, Grades 2 to 4 | 1 | 0
  Hypernatremia, Grades 3 to 4 | 0 | 0
  Hypoglycemia, Grades 1 to 4 | 22 | 4
  Hypoglycemia, Grades 2 to 4 | 2 | 1
  Hypoglycemia, Grades 3 to 4 | 0 | 0
  Hypokalemia, Grades 1 to 4 | 29 | 13
  Hypokalemia, Grades 2 to 4 | 1 | 1
  Hypokalemia, Grades 3 to 4 | 0 | 0
  Hyponatremia, Grades 1 to 4 | 55 | 15
  Hyponatremia, Grades 2 to 4 | 2 | 0
  Hyponatremia, Grades 3 to 4 | 0 | 0
  LDL cholesterol, Grades 1 to 4 | 107 | 22
  LDL cholesterol, Grades 2 to 4 | 46 | 10
  LDL cholesterol, Grades 3 to 4 | 15 | 3
  Lipase, Grades 1 to 4 | 67 | 7
  Lipase, Grades 2 to 4 | 35 | 3
  Lipase, Grades 3 to 4 | 12 | 0
  Total bilirubin, Grades 1 to 4 | 52 | 11
  Total bilirubin, Grades 2 to 4 | 42 | 10
  Total bilirubin, Grades 3 to 4 | 18 | 6
  Triglycerides, Grades 1 to 4 | 23 | 2
  Triglycerides, Grades 2 to 4 | 23 | 2
  Triglycerides, Grades 3 to 4 | 11 | 1
  Hemoglobin, Grades 1 to 4 | 11 | 6
  Hemoglobin, Grades 2 to 4 | 6 | 0
  Hemoglobin, Grades 3 to 4 | 2 | 0
  Neutrophils, Grades 1 to 4 | 37 | 9
  Neutrophils, Grades 2 to 4 | 14 | 4
  Neutrophils, Grades 3 to 4 | 7 | 2
  Platelets, Grades 1 to 4 | 22 | 7
  Platelets, Grades 2 to 4 | 11 | 1
  Platelets, Grades 3 to 4 | 4 | 0
  White Blood Cells, Grades 1 to 4 | 17 | 3
  White Blood Cells, Grades 2 to 4 | 7 | 1
  White Blood Cells, Grades 3 to 4 | 0 | 0

10. Secondary Outcome: DTG PK Parameters Including Maximum Plasma Drug Concentration (Cmax), Minimal Plasma Drug Concentration (Cmin), and Average Plasma Pre-dose Concentration (C0_avg)
Description: Cmax, Cmin and C0_avg were assessed by population pharmacokinetic (PK) modeling using sparse PK samples which were collected as follows: one pre-dose sample and one post-dose sample at 1 to 3 hours/4 to 12 hours at Week 4, one pre-dose sample at Week 24, and one pre-dose sample and one post-dose sample at 1 to 3 hours/4 to 12 hours at Week 48. Cmax, Cmin and C0_avg were estimated and reported here.
Time Frame: Pre-dose and at 1 to 3 hours or 4 to 12 hours post-dose at Week 4; Pre-dose at Week 24; Pre-dose and 1 to 3 hours or 4 to 12 hours post-dose at Week 48
Population: PK Concentration Population comprised of all participants who received DTG, underwent sparse PK sampling during the study, and provided evaluable DTG plasma concentration data. Only those participants with data available at the specified data points were assessed (represented by "n=X" in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | DTG 50 mg OD
Number analyzed (Participants) | 342
microgram/milliliter (µg/mL)
  C0_avg, n=342 | 0.926 (131)
  Cmax, n=340: number analyzed (Participants) | 340
  Cmax, n=340 | 3.21 (26.7)
  Cmin, n=340: number analyzed (Participants) | 340
  Cmin, n=340 | 0.849 (76.5)

11. Secondary Outcome: DTG PK Parameter Including Pre-dose Concentration (C0)
Description: C0 was assessed by population PK modeling using sparse PK samples which were collected as follows: one pre-dose sample and one post-dose sample at 1 to 3 hours/4 to 12 hours at Week 4, one pre-dose sample at Week 24, and one pre-dose sample and one post-dose sample at 1 to 3 hours/4 to 12 hours at Week 48. DTG predose concentration (C0) at Week 4, Week 24, and Week 48 was estimated and reported here.
Time Frame: Pre-dose at Weeks 4, 24 and 48
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | DTG 50 mg OD
Number analyzed (Participants) | 342
microgram/milliliter (µg/mL)
  Week 4, n=329: number analyzed (Participants) | 329
  Week 4, n=329 | 0.786 (143)
  Week 24, n=298: number analyzed (Participants) | 298
  Week 24, n=298 | 0.940 (132)
  Week 48, n=276: number analyzed (Participants) | 276
  Week 48, n=276 | 0.932 (152)

12. Secondary Outcome: DTG PK Parameters Including Area Under the Plasma Concentration-time Curve From Time Zero to Time Tau Over a Dosing Interval at Steady State (AUC[0-tau])
Description: AUC is defined as the area under the DTG concentration-time curve as a measure of drug exposure over time. AUC(0-tau) is defined as the area under the plasma concentration-time curve from time zero to time tau over a dosing interval at steady state, where tau is the length of the dosing interval of DTG. AUC was assessed by population pharmacokinetic (PK) modeling using sparse PK samples which were collected as follows: one pre-dose sample and one post-dose sample at 1 to 3 hours/4 to 12 hours at Week 4, one pre-dose sample at Week 24, and one pre-dose sample and one post-dose sample at 1 to 3 hours/4 to 12 hours at Week 48.
Time Frame: as for outcome 10
Population: PK Concentration Population: all participants who received DTG, underwent sparse PK sampling during the study, and provided evaluable DTG plasma concentration data. Only those participants available at the indicated time points were assessed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms*hour/milliliter (µg*hr/mL)
Arm/Group | DTG 50 mg OD
Number analyzed (Participants) | 340
Micrograms*hour/milliliter (µg*hr/mL) | 44.7 (40.5)

13. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-3 Levels (EQ-5D-3L) Utility Score
Description: The EQ-5D-3L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 3 levels for each dimension including 1=no problems, 2=some problems, 3=extreme problems. The health state is defined by combining the levels of answers from each of the 5 questions. Each health state is referred to in terms of a 5 digit code. Health state 5 digit code is translated into utility score, which is valued up to 1 (perfect health) with lower values meaning worse state. EQ-5D-3L utility score ranges from -0.594 to 1. Higher scores indicate better health. Baseline was the latest pre-dose assessment value (Day 1) and change from Baseline=post-dose value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: mITT-E Population. Only those participants with data available at the specified data points were assessed (represented by "n=X" in the category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Scores on a scale
  Week 24, n=350, 356: number analyzed (Participants) | 350 | 356
  Week 24, n=350, 356 | 0.010 (0.202) | 0.019 (0.204)
  Week 48, n=350, 356: number analyzed (Participants) | 350 | 356
  Week 48, n=350, 356 | 0.028 (0.179) | 0.013 (0.222)

14. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-3 Levels (EQ-5D-3L) Thermometer Scores
Description: The EQ-5D-3L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 3 levels for each dimension including 1=no problems, 2=some problems, 3=extreme problems. EQ-5D-3L included EQ visual Analogue scale (EQ VAS) 'Thermometer' which provided Self-rated current health status. Participants were asked to rate their current health status using the visual analogue scale 'Thermometer'. Score ranged from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores indicate better heath. Baseline was the latest pre-dose assessment value (Day 1) and change from Baseline=post-dose value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 354 | 361
Scores on a scale
  Week 24, n=350, 355: number analyzed (Participants) | 350 | 355
  Week 24, n=350, 355 | 6.800 (21.413) | 4.645 (18.279)
  Week 48, n=350, 355: number analyzed (Participants) | 350 | 355
  Week 48, n=350, 355 | 8.894 (20.356) | 5.597 (18.821)

15. Other Pre Specified Outcome: Absolute Values of Cluster of Differentiation 8+ (CD8+) Cell Counts at Weeks 4, 8, 12, 16, 24, 32, 40, and 48
Description: The absolute value data for CD8+ cell count was planned to be evaluated. The results for this outcome measure will never be posted.
Time Frame: At Weeks 4, 8, 12, 16, 24, 32, 40, and 48
Population: mITT-E Population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Change From Baseline in CD8+ Cell Counts at Weeks 4, 8, 12, 16, 24, 32, 40, and 48
Description: Change from Baseline data for CD8+ cell count was planned to be evaluated. The results for this outcome measure will never be posted.
Time Frame: Baseline (Day 1); Weeks 4, 8, 12, 16, 24, 32, 40, and 48
Population: as for outcome 15
Arm/Group | DTG 50 mg OD | RAL 400 mg BID
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs), non-serious AEs and all-cause mortality were collected from the start of study medication to the end of the study (up to Week 480)
Description: SAEs, non-serious AEs and all-cause mortality were collected in members of the Safety Population, comprised of all participants who received at least one dose of investigational product.
Groups:
- DTG~50mg QD: Participants received dolutegravir (DTG) 50 milligrams (mg) once daily (OD) + matching Raltegravir (RAL) placebo twice daily (BID), one in the morning (AM dose) and one in the evening (PM dose) + investigator selected background antiretroviral (ART) therapy for 48 weeks. Participants who successfully completed 48 weeks of treatment continued to have access to DTG in the Open-Label phase of the study.
- RAL~400mg BID: Participants received matching DTG placebo OD + RAL 400 mg BID as AM and PM doses + investigator selected background ART therapy for 48 weeks. Participants were discontinued from the study after completion of the Week 48 visit unless a participant successfully completed Week 48 and RAL was not approved and commercially available within the country, GSK continued to supply RAL in the Open-Label Phase until it was commercially available.
Arm/Group | DTG~50mg QD | RAL~400mg BID
All-Cause Mortality (participants affected / at risk) | 6/357 | 4/362
Serious Adverse Events (participants affected / at risk) | 73/357 | 46/362
Other Adverse Events (participants affected / at risk) | 250/357 | 206/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG~50mg QD (N=357) | RAL~400mg BID (N=362)
Pneumonia (Infections and infestations) | 7 (8) | 7 (7)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 2 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Coagulation factor deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Cytomegalovirus oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Extrapulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Histoplasmosis disseminated (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 (1) | 0 (0)
Immunoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infective myositis (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parvovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis liver (Infections and infestations) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Nasal valve collapse (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG~50mg QD (N=357) | RAL~400mg BID (N=362)
Diarrhoea (Gastrointestinal disorders) | 92 (134) | 64 (86)
Upper respiratory tract infection (Infections and infestations) | 72 (168) | 37 (82)
Headache (Nervous system disorders) | 43 (57) | 36 (41)
Nausea (Gastrointestinal disorders) | 35 (41) | 31 (38)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (61) | 26 (31)
Influenza (Infections and infestations) | 42 (69) | 34 (50)
Nasopharyngitis (Infections and infestations) | 43 (67) | 22 (23)
Urinary tract infection (Infections and infestations) | 35 (43) | 20 (24)
Vomiting (Gastrointestinal disorders) | 27 (32) | 20 (30)
Fatigue (General disorders) | 19 (21) | 26 (29)
Rash (Skin and subcutaneous tissue disorders) | 30 (34) | 21 (21)
Sinusitis (Infections and infestations) | 31 (41) | 17 (20)
Bronchitis (Infections and infestations) | 27 (45) | 15 (18)
Gastroenteritis (Infections and infestations) | 21 (22) | 7 (9)
Abdominal pain (Gastrointestinal disorders) | 21 (24) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 23 (25) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (38) | 27 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (37) | 16 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (25) | 20 (24)
Dizziness (Nervous system disorders) | 20 (21) | 13 (13)
Hypertension (Vascular disorders) | 39 (43) | 15 (16)
Depression (Psychiatric disorders) | 18 (19) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.